CLINICAL TRIAL: NCT07112170
Title: Consolidative Use of Radiotherapy to Block Oligoprogression in Patients With Metastatic Melanoma (CURB-Melanoma) - a Phase 2 Clinical Trial
Brief Title: Consolidative Use of Radiotherapy to Block Oligoprogression in Patients With Metastatic Melanoma
Acronym: CURB-Melanoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-5162
Record Dates: First submitted 2025-07-29; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Melanoma; OligoProgressive Metastatic Disease
Keywords: stereotactic body radiation therapy (SBRT); Melanoma
MeSH Terms: conditions — Melanoma | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): This is a single-arm trial, meaning all participants will receive the same treatment. There is no control or comparison group. All eligible patients will continue their existing first-line systemic therapy and receive additional radiation treatment-either stereotactic body radiotherapy (SBRT) or hypofractionated radiotherapy-directed at oligoprogressive lesions. The outcomes will be measured and analyzed based on this single group.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — SBRT will be delivered as per institutional standard.

SUMMARY:
This open-label, prospective, single-arm Phase II trial explores whether adding stereotactic body radiotherapy (SBRT) or hypofractionated radiotherapy to oligoprogressive lesions can help delay disease progression in patients with metastatic melanoma. Participants may have up to ten extracranial oligoprogressive sites, with no upper limit on the total number of metastatic lesions. The study aims to assess whether targeting these progressing sites with focused radiotherapy can extend progression-free survival in this patient population.

DETAILED DESCRIPTION:
his is an open-label, single-arm, Phase II study evaluating the use of stereotactic body radiotherapy (SBRT) or hypofractionated radiotherapy in patients with metastatic melanoma who have up to 10 extracranial oligoprogressive lesions while receiving first-line systemic therapy. Oligoprogression refers to progression at a limited number of sites, while the remaining disease remains controlled by systemic treatment.

Participants will continue their current systemic therapy and receive SBRT or hypofractionated radiotherapy to all oligoprogressive lesions. The study will assess whether this approach can delay overall disease progression and extend the duration of benefit from ongoing systemic therapy.

Imaging will be used to monitor disease progression, and blood samples will be collected at baseline, after radiation, and at disease progression for exploratory analysis. Additional outcomes include overall survival, time on current therapy, toxicity, quality of life, and out-of-field response.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* ECOG 0-2
* Willing and able to provide informed consent
* Metastatic melanoma detected on imaging and clinically confirmed.
* Treated with first line immunotherapy or BRAF inhibitors.
* No upper limit to the number of total metastatic sites, but a maximum of ten progressive metastatic sites, inclusive of primary disease and metastatic lesions, all of which must be extra cranial.
* Patients who had any prior radiation therapy near or overlapping with the oligoprogressive sites are allowed to enroll.
* All sites of oligoprogression that can be safely treated with SBRT or hypofractionated radiotherapy.

Exclusion Criteria:

* >10 extracranial sites of progressive disease.
* Pregnancy.
* Leptomeningeal disease.
* Serious medical comorbidities precluding radiotherapy, such as ataxia-telangiectasia or scleroderma.
* Prior radiotherapy near the oligoprogressive lesion precluding SBRT or hypofractionated radiotherapy due to exceeding OAR tolerance.
* Any psychological, sociological or geographical issue potentially hampering compliance with the study.
* Any other condition which in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2027-07-24 (Estimated); Study Completion 2028-07-24 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) assessed by radiological imaging using RECIST v1.1 criteria | From enrollment up to 24 months
  To determine if the addition of SBRT or hypofractionated radiation to progressive lesions improves progression-free survival in patients with metastatic melanoma.
  To determine if the addition of SBRT or hypofractionated radiation to progressive lesions improves progression-free survival in patients with metastatic melanoma. Radiological progression will be evaluated using CT, PET-CT, or MRI according to RECIST v1.1.

SECONDARY OUTCOMES:
Overall Survival (OS) measured from date of enrollment to death from any cause | Enrollment up to 24 months
Time on Current Systemic Therapy After Initial Oligoprogression | From enrollment up to 24 months
Out-of-field response assessed by radiological imaging (CT, PET-CT, or MRI) | From enrollment up to 24 months.
Toxicity assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | From start of SBRT through follow-up (up to 24 months)
Participant-reported adverse events measured using PRO-CTCAE questionnaire | From baseline through follow-up (up to 24 months)
Participant-reported quality of life measured using EORTC QLQ-C30 questionnaire | From baseline through follow-up (up to 24 months)

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No